CLINICAL TRIAL: NCT05774730
Title: Evaluation of the Effectiveness of Predicting the Integrity of Interlobar Fissures Based on Chest Image AI Technology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: 2022-NHLHCRF-LX-01-0202-2
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Emphysema quantitative analysis softwarebased on chest image AI technology
  Interventions: Other: Emphysema quantitative analysis software based on chest image AI technology
- artificial analysis
  Interventions: Other: artificial analysis of chest image
- imported Chartis detection system
  Interventions: Procedure: imported Chartis detection system

INTERVENTIONS:
Other: Emphysema quantitative analysis software based on chest image AI technology — The participants would undergo lung CT, and the integrity of interlobar fissure will be quantitatively analyses by software based on chest image AI technology.
  Groups: Emphysema quantitative analysis softwarebased on chest image AI technology
Other: artificial analysis of chest image — The participants would undergo lung CT, and the integrity of interlobar fissure will be artificially analyses.
  Groups: artificial analysis
Procedure: imported Chartis detection system — The participants would undergo imported Chartis detection system.
  Groups: imported Chartis detection system

SUMMARY:
The goal of observational study is to evaluate effectiveness of predicting the integrity of interlobar fissures based on chest image AI technology in patients with Chronic Obstructive Pulmonary Disease who will undergo lung volume reduction surgery with endobronchial valve implantation. The main question it aims to answer is: evaluation of the effectiveness of predicting the integrity of interlobar fissures based on chest image AI technology.

Participants will be evaluated by lung CT (quantitative analysis based on chest image AI technology and artificial analysis) and imported Chartis detection system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic obstructive pulmonary disease who meet the GOLD diagnostic criteria
* FEV1 ≤ 45% pred and FEV1/FVC<70%
* TLC>100% pred and RV>175% pred
* CAT≥18
* >50% of emphysema destruction
* Smoking prohibition>6 months
* Sign the informed consent form

Exclusion Criteria:

* PaCO2>8.0 kPa, or PaO2<6.0 kPa
* 6-minute walking test<160m
* Obvious chronic bronchitis, bronchiectasis or other infectious lung diseases
* Three hospitalizations due to pulmonary infection in the past 12 months before the baseline assessment
* Previous lobectomy, LVRS or lung transplantation
* LVEF<45% and or RVSP>50mmHg
* Anticoagulant therapy that cannot be stopped before surgery
* The patient has obvious immune deficiency
* Participated in other lung drug studies within 30 days before this study
* Pulmonary nodules requiring intervention
* Any disease or condition that interferes with the completion of the initial or subsequent assessment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic obstructive pulmonary diseases
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-26 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effect of lung volume reduction surgery | 1 month after bronchoscopic valve lung volume reduction
  Lung CT
Therapeutic effect of lung volume reduction surgery | 3 months after bronchoscopic valve lung volume reduction
  Lung CT
Therapeutic effect of lung volume reduction surgery | 6 months after bronchoscopic valve lung volume reduction
  Lung CT
the integrity of interlobar fissure | Before bronchoscopic valve lung volume reduction
  Emphysema quantitative analysis softwarebased on chest image AI technology, artificial analysis and imported Chartis detection system